CLINICAL TRIAL: NCT06364904
Title: A Multicenter, III Stage, Randomized Controlled Trail on the Safety and Efficacy of the Combination of Tislelizumab With Cisplatin and Gemcitabine, With or Without Trilaciclib in Untreated Unresectable and Metastatic Urothelial Carcinoma.
Brief Title: A Clinical Trail to Determine the Safety and Efficacy of the Combination of Tislelizumab With Cisplatin and Gemcitabine, With or Without Trilaciclib for Patients With Untreated Unresectable and Metastatic Urothelial Carcinoma.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-123-02
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Bladder Cancer
Keywords: Immune Checkpoint Inhibitor; CDK4/6 Inhibitor; Cisplatin; Tislelizumab; Gemcitabine; Trilaciclib
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — tislelizumab; Cisplatin; Gemcitabine; trilaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gemcitabine plus Cisplatin (Active Comparator): During each 21 days study cycle(up to 6 cycles), all participants will receive:
  1. Tislelizumab: Taken 1x time at d1 each cycle or until it is determined participant must stop the drug.
  2. Gemcitabine: d1, d8 each cycle or until it is determined participant must stop the drug.
  3. Cisplatin: d2 each cycle or until it is determined participant must stop the drug.
  Tislelizumab maintenance therapy:after chemoimmunotherapy, q3W until it is determined participant must stop the drug, or 2 years of treatment is completed.
  Interventions: Drug: Tislelizumab, Cisplatin, Gemcitabine
- Gemcitabine, Cisplatin plus Trilaciclib (Experimental): During each 21 days study cycle(up to 6 cycles), all participants will receive:
  1. Tislelizumab: Taken 1x time at d1 each cycle or until it is determined participant must stop the drug.
  2. Gemcitabine: d1, d8 each cycle or until it is determined participant must stop the drug.
  3. Cisplatin: d2 each cycle or until it is determined participant must stop the drug.
  4. Trilaciclib: d1, d2, d8 each cycle or until it is determined participant must stop the drug.
  Tislelizumab maintenance therapy:after chemoimmunotherapy, q3W until it is determined participant must stop the drug, or 2 years of treatment is completed.
  Interventions: Drug: Tislelizumab, Cisplatin, Gemcitabine and Trilaciclib

INTERVENTIONS:
Drug: Tislelizumab, Cisplatin, Gemcitabine and Trilaciclib — Chemoimmunotherapy:
  1. Tislelizumab: 200mg, 1x time at d1 each cycle
  2. Gemcitabine: 1000mg/ m2, in d1, d8 each cycle
  3. Cisplatin: 70 mg/m2, in d2 each cycle
  4. Trilaciclib: 240mg/m2, d1, d2, d8 each cycle
  Tislelizumab maintenance therapy: after chemoimmunotherapy, 200mg, q3W.
  Arms: Gemcitabine, Cisplatin plus Trilaciclib
Drug: Tislelizumab, Cisplatin, Gemcitabine — Chemoimmunotherapy:
  1. Tislelizumab: 200mg, 1x time at d1 each cycle
  2. Gemcitabine: 1000mg/ m2, in d1, d8 each cycle
  3. Cisplatin: 70 mg/m2, in d2 each cycle
  Tislelizumab maintenance therapy: after chemoimmunotherapy, 200mg, q3W.
  Arms: Gemcitabine plus Cisplatin

SUMMARY:
The aim of this study is to see whether the Trilaciclib is safe and effective in slowing down the growth of bladder cancer in patients while taking chemoimmunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study, able to provide written informed consent and can understand and agree to comply with the requirements of the study and schedule of assessments.
2. Participants diagnosed histologically or cytologically with locally advanced or metastatic urothelial carcinoma (UC) of the renal pelvis, ureter, bladder, or urethra. Eligible subjects for inclusion are those with a mixed histologic type, as assessed by the investigator, with urothelial component >50% and plasmacytoid subtype <10%. Patients with histologically confirmed and radiologically assessed locally advanced or metastatic urothelial carcinoma of the urinary tract.
3. Participants judged by the investigator to be tolerant of platinum-based therapy. Participants intolerant to platinum chemotherapy must meet at least one of the following criteria: ECOG performance status >1 or Karnofsky performance status 60% to 70%; creatinine clearance less than 60 ml/min; hearing loss ≥ Grade 2 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5; peripheral neuropathy ≥ Grade 2 according to NCI-CTCAE version 5; New York Heart Association Class III or IV heart failure.
4. Must provide surgical or biopsy tumor tissue samples, and concurrent submission of relevant pathology reports is required. Participants are able to submit fresh surgical tissue or submit pathology slides for examination.
5. ECOG Performance Status 0 or 1
6. The participants must have well-functioning organ systems, as measured by the following screening laboratory values (obtained within ≤14 days before enrollment):

   a. When screening for the following parameters, participants must not have used growth factor support within ≤14 days before sample collection: i. Neutrophil absolute count ≥ 1.5x10^9/L ii. Platelets ≥ 90x10^9/L iii. Hemoglobin ≥ 90g/L b. International normalized ratio or activated partial thromboplastin time ≤ 1.5 times the upper limit of normal (ULN) c. Calculated creatinine clearance ≥ 50 mL/min d. Serum total bilirubin ≤ 1.5×ULN (if Gilbert's syndrome or indirect bilirubin concentration indicates extrahepatic elevation, should be ≤ 3×ULN) e. AST, ALT, and alkaline phosphatase ≤ 2.5×ULN
7. Women who are not pregnant or not of childbearing potential must be willing to use effective contraception during the study and for ≥120 days after the last dose of toripalimab monotherapy or chemotherapy (whichever occurs later). Additionally, they must have a negative urine or serum pregnancy test result within ≤7 days before enrollment. Non-sterilized men must be willing to use effective contraception during the study and for ≥120 days after the last dose of toripalimab monotherapy or chemotherapy (whichever occurs later).
8. According to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, at least one participant with measurable lesions is required.
9. Participants with an expected survival of ≥3 months.

Exclusion Criteria:

1. Known active or untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. For patients with previously treated brain metastases, enrollment is not allowed if there has been CNS disease stability for at least 4 weeks before the first dose of study treatment and discontinuation of corticosteroid therapy for brain metastases for at least 2 weeks before the start of study treatment.
2. Prior treatment with therapies targeting PD-1, PD-L1, PD-L2, CTLA-4, or other agents specifically targeting T-cell co-stimulation or checkpoint pathways.
3. Receipt of other approved systemic anticancer therapy or systemic immunomodulatory agents (including but not limited to interferons, interleukins, and tumor necrosis factor) within 28 days before enrollment.
4. Prior radiotherapy for bladder cancer.
5. Prior systemic treatment for tumors, except:

   1. For patients previously treated with systemic chemotherapy, a treatment-free interval of at least 12 months from the last treatment to the start of drug treatment.
   2. Local intravesical chemotherapy or immunotherapy, completed at least 1 week before the start of study treatment.
6. Major surgery or significant trauma within 28 days before enrollment (placement of vascular access device and transurethral resection of bladder tumor [TURBT] are not considered major surgery).
7. Severe chronic or active infection requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days before enrollment (HBV infection is excluded according to exclusion criterion 11).
8. Receipt of live vaccines within 28 days before enrollment (seasonal injections of influenza vaccine are usually inactivated vaccines and are allowed. Nasal vaccines are live vaccines and are not allowed).
9. Active autoimmune diseases requiring systemic treatment, as determined by the investigator, which could affect the safety of study treatment.
10. Long-term use of high-dose steroids or other immunosuppressive agents, as determined by the investigator, which could affect the safety of study treatment.
11. Known potassium, sodium, calcium abnormalities, or hypoalbuminemia, interstitial lung disease, non-infectious pneumonia, or other uncontrolled systemic diseases, including diabetes, hypertension, cardiovascular diseases (e.g., active cardiac disease within 6 months before enrollment, including severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, and requiring medication for ventricular arrhythmias).
12. Untreated chronic hepatitis B patients with HBV DNA ≥500 IU/mL (2500 copies/mL) or HBV carriers are not eligible. Note: Patients with inactive hepatitis B surface antigen carriers or stable active HBV infection (HBV DNA <500 IU/mL [2500 copies/mL]) after continuous antiviral treatment can be enrolled. HBV DNA testing is performed only in patients positive for antibodies to the hepatitis B core antigen.
13. Patients with active hepatitis C are not eligible. Patients who test negative for HCV antibodies during the screening period or, if positive, test negative for HCV RNA after positive HCV antibody testing can be enrolled. Only patients positive for HCV antibodies need HCV RNA testing.
14. History of immune deficiency (including human immunodeficiency virus [HIV] positive, other acquired, congenital immunodeficiency diseases) or a history of allogeneic stem cell transplantation or organ transplantation.
15. Known allergies to other monoclonal antibodies.
16. Known allergies to any study drug or excipient.
17. Patients with toxic side effects (due to any treatment) that have not returned to baseline or a stable level, unless the investigator does not believe that such toxic side effects may pose a safety risk (e.g., hair loss, neurologic symptoms, and specific laboratory abnormalities).
18. Underlying medical conditions, alcohol/drug abuse, or dependence that may adversely affect the administration of study drug, interpretation of results, or lead to a high risk of treatment complications.
19. Concurrent participation in another therapeutic clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Progression-Free Survival(PFS) | 24 months
  Progression free survival was determined from start date of treatment to date of progression for patients who progressed or date of death for patients who died without progressing. The observations of patients remaining alive and progression free were censored at the date of last disease evaluation. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Percentage of Participants With Incidence of Grade 3/4 Neutropenia | Within 28 days of initial dosing
  The proportion of participant with neutrophils with values < 1*10^9/L during treatment.

SECONDARY OUTCOMES:
Rate of ORR | 60 months
  The responses rate (PR+CR) in participants based on imaging [CT scan of chest, abdomen, and pelvis (or MRI of abdomen and pelvis with CT chest without contrast when appropriate)]
overall survival (OS) | 60 months
  OS was measured from the date the participant started study to death for any reason.
Safety and AE | 60 months
  Number of unique patients who had a treatment-related (possible, probable, or definite) adverse event using the Medical Dictionary for Regulatory Activities (MedDRA) terms and graded per NCI-CTCAE v5.0.
  Number and Grade of patients who had a surgery-related adverse event (surgery-related AE) will be measured according to the Clavien-Dindo classification.
Disease Control Rate(DCR) | 60 months
  The responses rate (PR+CR+SD) in participants based on imaging [CT scan of chest, abdomen, and pelvis (or MRI of abdomen and pelvis with CT chest without contrast when appropriate)].
During Of Response(DOR) | 60 months
  During Of Response(DOR) was measured from the date from the first evaluation of the tumor as CR or PR to the first evaluation as PD or death from any cause.
Biomarker Endpoint Analyses | 60 months
  Patients' biomarkers in urine, blood, and tumor tissues (include CPS, TPS, TMB, Ki67, etc.) will be detected with the treatment of the combination of Tislelizumab with Cisplatin and Gemcitabine, with or without Trilaciclib in untreated unresectable and metastatic urothelial.

CONTACTS AND LOCATIONS:
Overall Officials: Tianxin Lin, Ph.D, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (8):
- China (8):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan